CLINICAL TRIAL: NCT03889119
Title: Stereotactic Body Radiation Therapy (SBRT) for the Management of Carcinoma of the Prostate: Quality of Life Data After Primary Stereotactic Body Radiation Therapy for Localized Prostate Cancer
Brief Title: Stereotactic Body Radiation Therapy (SBRT) for Prostate Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hoag Memorial Hospital Presbyterian (Other)
Responsible Party: Principal Investigator, Kevin Lin, Radiation Oncologist, Hoag Memorial Hospital Presbyterian
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 115-16-CA
Record Dates: First submitted 2019-03-19; First posted 2019-03-26 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery; Radiation

STUDY DESIGN:
Intervention Model Description: SBRT for the management of localized prostate cancer is a Phase II non-randomized clinical trial open to patients with biopsy proven localized prostate cancer. Patients will be deemed eligible for SBRT in any risk group categorization based upon the standard D'Amico stratification:
  * Low-risk: initial PSA <10 and clinical stage T1c-T2a/b and biopsy Gleason grade 3+3
  * Intermediate-risk: initial PSA >10 but <20 or clinical stage T2c or biopsy Gleason grade 3+4 or 4+3
  * High-risk: initial PSA >20 or clinical stage T3 or biopsy Gleason grade 4+4 or higher).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Elekta Versa HD (Active Comparator): This study seeks to investigate biochemical failure rates for patients treated with SBRT utilizing Elekta machines, as well as obtain quality of life data and assess the intrafraction motion in approximately 15 patients for 5 years following SBRT.
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT) radiation for prostate cancer utilizing the Elekta Versa or Agility System.
- Agility Systems (Other): This study seeks to investigate biochemical failure rates for patients treated with SBRT utilizing Agility Systems, as well as obtain quality of life data and assess the intrafraction motion in approximately 15 patients for 5 years following SBRT.
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT) radiation for prostate cancer utilizing the Elekta Versa or Agility System.

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy (SBRT) radiation for prostate cancer utilizing the Elekta Versa or Agility System. — SBRT uses advanced imaging techniques to deliver targeted radiation to a tumor. The Elekta Versa and Agility Systems are approved by the Food and Drug Association (FDA) for SBRT treatment of cancer.
  Other Names: Cyberknife

SUMMARY:
The purpose of this study is to learn the long term efficacy and side effects associated with utilizing Stereotactic Body Radiation Therapy (SBRT) radiation for prostate cancer utilizing the Elekta Versa or Agility System. SBRT uses advanced imaging techniques to deliver targeted radiation to a tumor. The Elekta Versa and Agility Systems are approved by the Food and Drug Association (FDA) for SBRT treatment of cancer.

Traditional External beam radiation therapy (EBRT) for prostate carcinoma is typically done over the course of approximately 42-45 daily treatments SBRT is a way to condense this treatment into a course of 5 treatments, delivering more dose per day.

DETAILED DESCRIPTION:
Prostate cancer is the most common cancer diagnosed in men, and ranks second in estimated deaths. The current standard of care for localized prostate cancer consists of observation, surgery or radiation therapy. From a radiation perspective, accepted options include external beam radiation therapy, brachytherapy, or a combination of those. Acceptable external beam radiation options are further defined as conventionally fractionated (over approximately 8-9 weeks), or moderately hypo-fractionated (over approximately 4-6 weeks).

Stereotactic body radiation therapy (SBRT) is a newer technique, allowing treatment to be delivered in an extremely hypo-fractionated regimen (i.e. in 5 fractions). Current consensus guidelines describe SBRT as "a cautious alternative to conventionally fractionated regimens at clinics with appropriate technology, physics, and clinical expertise."

The goal of any therapy is to maximize the effect of that treatment on cancer cells and minimize any effect on normal tissue. In radiation therapy, this is mainly done through dose targeting (i.e. limiting the radiation dose to the targets and minimizing dose to normal surrounding organs). Advancements in radiation therapy have allowed for better targeting, resulting in shrinking margins of treatment around cancer cells.

The therapeutic window can also be optimized through the use of fractionation (i.e. amount of dose delivered per day) in radiation therapy. Since cancerous and normal tissue cells respond differently to changes in fractionation, the therapeutic window could theoretically be improved by choosing a fractionation pattern to which cancer cells are more sensitive. Historical generalizations put cancer cells into the category of early responding tissues, which would make them more sensitive to cell death when radiation is delivered in a protracted fractionation pattern, such as over 8-9 weeks of radiation therapy.

However, studies have emerged which suggest that prostate cancer is unlike other cancers and reactive more like late responding tissues. With that in mind, prostate cancer cells could be more sensitive to high doses per fraction, which could provide a radiobiological advantage and a greater therapeutic window with the use of SBRT.

Very promising early results utilizing SBRT for prostate cancer treatment have been described in the literature, and multiple ongoing phase 3 trials are underway.

Aside from a potential therapeutic advantage, SBRT also offers a more cost effective solution to patients with prostate cancer, with less impact on their daily lives (only needing to come in for 5 treatments instead of 40-45 treatments).

Much of the literature on SBRT has been done utilizing the CyberKnife system. But the Elekta Versa HD and Agility Systems available at Hoag provides a unique opportunity for faster treatment delivery and 4D imaging during treatment. The Elekta Versa HD and Agility systems are approved by the FDA for SBRT treatment of cancer.

This study seeks to investigate biochemical failure rates for patients treated with SBRT utilizing Elekta machines, as well as obtain quality of life data and assess the intrafraction motion in approximately 15 patients for 5 years following SBRT.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of adenocarcinoma of the prostate History/physical examination with digital rectal examination of the prostate
* Histological evaluation of prostate biopsy with assignment of Gleason score to the biopsy material.
* Clinical stage T1-3 (AJCC 7th edition).
* Males age ≥ 18
* Patient must be able to provide study-specific informed consent prior to study entry.
* Willingness and ability to complete the Expanded Prostate Cancer Index Composite (EPIC) questionnaire

Exclusion Criteria:

* Evidence of distant metastases
* Regional lymph node involvement
* Previous radical surgery (prostatectomy), cryosurgery, or HIFU for prostate cancer
* Previous pelvic irradiation, prostate brachytherapy
* Previous or concurrent cytotoxic chemotherapy for prostate cancer

There are no exclusions due to co-morbid disease or illnesses except for patients with severe inflammatory bowel disease

No life expectancy restrictions will apply

Performance Status will not be considered

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is open to patients with a pathologic diagnosis of localized prostate cancer and have expressed a desire to receive SBRT over other therapies
Enrollment: 100 (Estimated)
Dates: Start 2016-10-21 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary aim of this study is to examine biochemical failure rates after SBRT for patients with low, intermediate, and high risk localized non-metastatic prostate cancer. | 5 years
  The number of patients demonstrating biochemical failure will be assessed. Biochemical failure will be defined using the Phoenix definition (Roach et al. IJROBP 2006), which is defined as a rise above nadir PSA + 2 ng/ml.

SECONDARY OUTCOMES:
The secondary aim is to obtain quality of life data to examine the potential complications associated with SBRT: detailed symptom questionnaire | 5 years
  Expanded Prostate Cancer Index Composite for Clinical Practice (EPIC-CP) (Chang J Urol 2011) total symptom score change from baseline will be assessed. This total score ranges from 0-60, with higher scores representing more symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Hoag Memorial Hospital Presbyterian, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No